CLINICAL TRIAL: NCT02656810
Title: A Double-Masked, Randomized, Two-Treatment Cross-over Study Comparing the Pharmacokinetics of PF708 and Forteo Administered by Subcutaneous Injection in Healthy Adult Subjects
Brief Title: A Comparison Study of PF708 and Forteo in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfenex, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PF708-101
Record Dates: First submitted 2016-01-12; First posted 2016-01-15 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A (Experimental): Single subcutaneous injection of two teriparatide products (PF708 and Forteo)
  Interventions: Drug: Teriparatide
- Sequence B (Experimental): Single subcutaneous injection of two teriparatide products (Forteo and PF708)
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Teriparatide — Single subcutaneous injection
  Other Names: PF708

SUMMARY:
The purpose of this study is to compare the pharmacokinetics (blood levels) of two teriparatide products, PF708 and Forteo, in healthy subjects.

DETAILED DESCRIPTION:
This is a double-masked, randomized, two-treatment cross-over study in healthy adult subjects. Half of the subjects will be randomized to receive PF708 first and Forteo second (Sequence A), and the other half will be randomized to receive the drugs in reverse sequence (Sequence B),

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-50 years at the time of Informed Consent.
* Able to understand and sign the written Informed Consent Form (ICF).

Exclusion Criteria:

* History of or positive test result for human immunodeficiency virus (HIV), hepatitis C virus [test for hepatitis C virus antibody (HCV Ab)] or hepatitis B virus [test for hepatitis B surface antigen (HBsAg)].
* Female subjects who are pregnant or have a positive pregnancy test result, currently breastfeeding, or planning to become pregnant during the course of the study.
* Blood donation (greater than or equal to 500 mL) within 30 days prior to screening.
* History of Paget's disease of bone.
* History of prior external beam or implant radiation therapy involving the skeleton.
* Active urolithiasis or primary hyperparathyroidism.
* History of alcohol or substance abuse within 3 years prior to screening.
* Previous treatment, including for investigational purposes, with any products (e.g., Forteo, Natpara) derived from human parathyroid hormone (PTH).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Serum area-under-the-curve (AUC) of PF708 and Forteo | 24 hours
Serum maximum concentration (Cmax) of PF708 and Forteo | 24 hours

SECONDARY OUTCOMES:
Change in serum calcium concentration after a single subcutaneous dose of PF708 and Forteo | 0-24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hubert C Chen, M.D., Study Director — Pfenex, Inc
Locations (1):
- Covance Clinical Research Unit, Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided